CLINICAL TRIAL: NCT02436408
Title: VISmodegib for ORbital and Periocular Basal Cell Carcinoma (VISORB)
Brief Title: VISmodegib for ORbital and Periocular Basal Cell Carcinoma
Acronym: VISORB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.022; HUM00082579 (Other: University of Michigan)
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vismodegib (Experimental): 150mg taken orally once daily
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib

SUMMARY:
Basal cell carcinoma (BCCA) is the most common human cancer, and frequently affects facial structures. While rarely fatal, facial BCCA can be disfiguring and expensive to treat.

Vismodegib is a small molecule inhibitor of SMO developed for the treatment of tumors in which the Hh signaling pathway appears to contribute to the development and maintenance of tumorigenesis. Vismodegib was recently approved by the Food and Drug Administration (FDA) for treatment of metastatic and locally advanced BCCA. Recent reports have suggested that vismodegib treatment for orbital BCCA may facilitate eye preservation even if surgery is eventually required

In order to assess the potential of vismodegib to improve the ophthalmic outcomes following treatment for orbital and/or periocular BCCA, this study will follow patients with globe-threatening orbital and lacrimal-threatening periocular BCCA who are being treated with vismodegib as standard of care.

Patients with tumors that do not respond to treatment with Vismodegib, and those who have a good response but poor tolerance of Vismodegib, will be offered surgical excision of the tumor. Patients with a good response and good tolerance of Vismodegib may continue the treatment as long as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age with locally advanced or recurrent orbital or periorbital basal cell carcinoma (BCCA), or a medial canthal BCCA that threatens the lacrimal drainage system.
* Clinical assessment score obtained at baseline.
* Medical Oncology screening performed at baseline.
* Adequate BCCA size and location.
* Adequate hematopoietic capacity, hepatic and renal function.
* Male patients must agree to use condoms during treatment and for 3 months after last dose.
* Male patients must agree to not donate sperm during treatment and for 3 months after last dose.
* Participant must agree not to donate blood during the study and for 7 months after last dose.
* Informed consent signed.
* If the patient consents to enroll, then blood will be drawn and stored for biomarker analysis.

Exclusion Criteria:

* Inability or unwillingness to swallow capsules.
* Inability or unwillingness to comply with study procedures.
* Pregnant, lactating, or breast feeding women.
* Women of childbearing potential.
* Uncontrolled medical illness.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Age under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cagri Besirli, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Unsworth SP, Tingle CF, Heisel CJ, Eton EA, Andrews CA, Chan MP, Bresler SC, Kahana A. Analysis of residual disease in periocular basal cell carcinoma following hedgehog pathway inhibition: Follow up to the VISORB trial. PLoS One. 2022 Dec 1;17(12):e0265212. doi: 10.1371/journal.pone.0265212. eCollection 2022. PMID 36455049
- [Derived] Kahana A, Unsworth SP, Andrews CA, Chan MP, Bresler SC, Bichakjian CK, Durham AB, Demirci H, Elner VM, Nelson CC, Kim DS, Joseph SS, Swiecicki PL, Worden FP. Vismodegib for Preservation of Visual Function in Patients with Advanced Periocular Basal Cell Carcinoma: The VISORB Trial. Oncologist. 2021 Jul;26(7):e1240-e1249. doi: 10.1002/onco.13820. Epub 2021 May 31. PMID 33988881
- [Derived] Rao RC, Chan MP, Andrews CA, Kahana A. EZH2, Proliferation Rate, and Aggressive Tumor Subtypes in Cutaneous Basal Cell Carcinoma. JAMA Oncol. 2016 Jul 1;2(7):962-3. doi: 10.1001/jamaoncol.2016.0021. No abstract available. PMID 27054919

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vismodegib
Started | 35
Completed | 34
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vismodegib
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 69 [45 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With a Score of 21 or Greater by the Visual Assessment Weighted Score (VAWS).
Description: The VAWS was developed for the purpose of this study. It is made up of standard ophthalmic exam points, as well as subjective assessment of tearing and overall patient satisfaction. The maximum score is 50 and a score of 21 or greater will be considered a good outcome.
Time Frame: Until end of study treatment (up to 15 months after start of study treatment); treatment duration ranged from 53 - 386 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 34
Participants | 34

2. Secondary Outcome: Number of Patients With Progressive Disease (PD)
Description: Treatment response will be determined per Response Evaluation Criteria in Solid Tumors (RECIST) protocol, using clinical measurements and/or tumor imaging measurements (determined by treating physician).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 34
Participants | 0

3. Secondary Outcome: Number of Patients With a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) AND Good Tolerance of Vismodegib
Description: Tolerance will be self-reported by patient. Treatment response will be determined per Response Evaluation Criteria in Solid Tumors (RECIST) protocol, using clinical measurements and/or tumor imaging measurements (determined by treating physician).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 34
Participants | 7

4. Secondary Outcome: Number of Patients With a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) AND Poor Tolerance of Vismodegib
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 34
Participants | 27

ADVERSE EVENTS:
Time Frame: Up to 15 months after start of study treatment; data was collected on study for 62 months total
Arm/Group | Vismodegib
All-Cause Mortality (participants affected / at risk) | 2/35
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib (N=35)
Acute coronary syndrome (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Heart failure (Cardiac disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Vascular disorders - Other (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vismodegib (N=35)
Anemia (Blood and lymphatic system disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Cataract (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 8
Eye pain (Eye disorders) | 1
Eyelid function disorder (Eye disorders) | 3
Watering eyes (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Edema face (General disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 12
Fever (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 1
Pain (General disorders) | 4
Papulopustular rash (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Weight loss (Investigations) | 12
Anorexia (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 26
Facial muscle weakness (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Spasticity (Nervous system disorders) | 7
Agitation (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Libido decreased (Psychiatric disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 17
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The initial study design aimed to enroll 50 patients; however, the study was terminated early as a consequence of the therapeutic and administrative challenges posed by the novel coronavirus pandemic and because the interim analysis revealed that the study at the point of termination was sufficient to achieve statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02436408/Prot_SAP_000.pdf